CLINICAL TRIAL: NCT02568085
Title: Randomized Controlled Trial Evaluating Use of Arista Absorbable Surgical Hemostatic Powder in Total Thyroidectomy With and Without Neck Dissections
Brief Title: Trial Evaluating Use of Arista in Total Thyroidectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Arista for Thyroids
Record Dates: First submitted 2015-09-29; First posted 2015-10-05 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Thyroidectomy; Seroma
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): thyroidectomy + Arista
  Interventions: Device: Arista
- 2 (No Intervention): Thyroidectomy
- 3 (Experimental): Thyroidectomy with neck + Arista
  Interventions: Device: Arista
- 4 (No Intervention): Thyroidectomy with neck

INTERVENTIONS:
Device: Arista — Arista™ AH is a medical device intended for application to surgical wound sites as an absorbable hemostat. The device is a fine, dry, sterilized white powder that is biocompatible, non-pyrogenic, and is typically absorbed within 24 to 48 hours.
  Arms: 1; 3

SUMMARY:
This is a single-blinded randomized controlled trial to evaluate the effectiveness of Arista hemostatic matrix powder (Arista® AH, C. R. Bard, Inc. Davol, Warwick, RI) in reducing drainage output after total thyroidectomy with and without lateral neck dissections. Increased drainage in total thyroidectomy and neck dissection wound beds can lead to seroma formation with possible secondary infection, delayed hospital discharge, and additional home care needs for drain care. Arista is an inert plant based absorbable surgical hemostatic powder that can be easily applied to broad surgical fields to reduce bleeding and seroma rates. Therefore, its application to thyroidectomy and neck dissection wound beds may bear significant potential benefit.

DETAILED DESCRIPTION:
This is a single-blinded randomized controlled trial to evaluate the effectiveness of Arista hemostatic matrix powder in reducing drainage output after total thyroidectomy with and without lateral neck dissections. Increased drainage in total thyroidectomy and neck dissection wound beds can lead to seroma formation with possible secondary infection, delayed hospital discharge, and additional home care needs for drain care. Arista is an inert plant based absorbable surgical hemostatic powder that can be easily applied to broad surgical fields to reduce bleeding and seroma rates. Therefore, its application to thyroidectomy and neck dissection wound beds may bear significant potential benefit.

Specific Aim 1: The main hypothesis of the study is that the use of Arista in total thyroidectomy with and without lateral neck dissections prior to closure will reduce postoperative drain outputs and time to drain removal compared to total thyroidectomy with and without lateral neck dissection closed without Arista.

Specific Aim 2: This study will also evaluate the secondary hypotheses that Arista will reduce postoperative hematoma and seroma rates and hospital length of stay in total thyroidectomies with and without lateral neck dissections.

INTRODUCTION

Total thyroidectomy is an increasingly common procedure performed where the entire thyroid gland is removed for either benign or malignant disease. Common indications include multinodular goiter, Graves disease, and thyroid carcinoma. Between 2006 and 2011 the number of total thyroidectomies performed in the United States increased by 12% per year, from 45,558 to 72,344 according the to the American Cancer Society. In 2011 48,000 total thyroidectomies were performed for malignant disease which often requires additional lateral neck dissection.

Although patients do very well after total thyroidectomy with over 90% 5-year survival for patients with well-differentiated thyroid carcinoma, total thyroidectomy with and without lateral neck dissection still carries the potential for serious complications including neck hematomas or seromas. Postoperative fluid collections continue to be problematic after thyroidectomy with or without lateral neck dissection with hematoma rates of 1-3% and seroma rates of 4-7%. In order to try and reduce the rate of hematomas and seromas after total thyroidectomy with or without lateral neck dissection, the majority of surgeons place closed suction drains (CSDs) in the wound prior to closure. Surgeons generally use drains in an attempt to identify, reduce, and or prevent hematomas and seromas even though there is little evidence to support this practice.

At this institution, it is common practice to place single drain in the thyroid bed and another drain in the neck of a lateral neck dissection is preformed and only remove drains once the output is less than 30ml over a 24-hour period or 15ml over a 12-hour period with a downward trend. Meeting this output volume criterion often takes several days. Often, a patient will be given the decision to be discharged home with a drain or wait and continue inpatient hospitalization until drain output requirements are met. Prolonged drain can lead to increased infection risks and unnecessary hospital stay. According the Healthcare Cost and Utilization Project, an average inpatient hospitalization in 2009 cost $2,000 per day, and is increasing. The reduction of an average of just one hospital day per thyroidectomy patient could potential save $144,688,000 dollars a year. An evaluation of Arista use on reducing drain output may reveal unnecessary expenses related to increased hospital length of stay and could lead to significant cost savings. Further, the associated morbidity and health care costs of potential seroma or infected seroma complications may be avoided.

According to the manufacturer, Arista uses Microporous Polysaccharide Hemospheres (MPH) technology to catalyze the clotting cascade and effectively dehydrate tissue to initiate hemostasis in broad areas. Major advantages of Arista are that it has been shown to be safe and effective across multiple surgical disciplines, is completely absorbed in 24-48 hours, and contains no human or animal components.

Previous works support the idea that Arista could be effective in reducing postoperative fluid collection and drainage time in free flap donor sites. However, this would be a new application of Arista with wide applicability that has not been previously described.

Possible Influence On Clinical Practice

Total thyroidectomies with and without lateral neck dissections, and surgery in general, have evolved in an era of increased attention to quality of life and cost savings. The most radical neck dissections are increasingly being replaced by more focused "functional" and "selective" neck dissections, during which the spinal accessory nerve, sternocleidomastoid muscle, internal jugular vein, and cervical sensory nerves are preserved and a more narrowly defined set of lymph node levels are excised, based on oncologic risk profiling. Finding Arista can decrease total thyroidectomy with or without lateral neck dissection drain output and lead to earlier drain removal could improve the quality of life of patients, significantly decrease the cost of care, and potentially decrease drain-associated infections.

This study seeks to critically evaluate current clinical practice paradigms to better understand the potential benefit of Arista post thyroidectomy with or without lateral neck dissection wound beds. A prospective, randomized, controlled, single-blinded trial is the clearest methodology to evaluate the possible by limiting bias and confounding variables. No clinical trial of this level has been performed on this topic; thus, this proposal is novel and the findings of the study are potentially important.

SUBJECTS AND METHODS

Patient Population and Enrollment

All adult patients (18 years old and over) undergoing total thyroidectomy with or without lateral neck dissection by one of two Head and Neck Surgery faculty members at UCSF will be included in enrollment for the study and consecutively registered.

Exclusion criteria will consist of patient age under 18, requirement of postoperative anticoagulant medications other than routine deep venous thrombosis prophylaxis (such as warfarin), and presence of clotting or bleeding disorder.

Study Protocols and Surgical Description

If successfully enrolled to the study, a randomized packet containing the patient's research ID number will be pulled and included into the patient's chart. Randomization will be done at the initiation of the study by creating a randomization list with blocking and stratification by surgeon. An envelope containing the patients randomized group assignment will not be opened until the end of the procedure just prior to closure.

The patients will be randomized to one of four groups. Groups 1 and 2 will consist of patients undergoing total thyroidectomy with possible central neck dissection but not lateral neck dissection. Patients in Group 1 will have 3 grams of Arista applied diffusely to the wound bed before primary closure. Patients in Group 2 will not have any Arista applied. Per routine, patients in both groups will have a single 10 French Jackson-Pratt drain will be placed within the thyroid bed and removed per a standardized protocol.

Groups 3 and 4 will consist of patients undergoing total thyroidectomy with lateral neck dissection. Patients in Group 3 will have 3 grams of Arista applied diffusely to the thyroid and neck wound bed before primary closure. Patients in Group 4 will not have any Arista applied. All incisions will be closed in 3 layers with 3-0 vicryl, 4-0 monocryl, and 5-0 fast absorbing sutures. All patients will receive standardized postoperative orders including inpatient antibiotics not to exceed 24hrs (unless an infection is suspected) and DVT prophylaxis; either weight based subcutaneous heparin or enoxaparin.

The drain will only be removed once output is less than 30ml per 24hr or 15ml per 12hr with downward trend. All patients will receive similar postoperative instructions including wound care, with and without drain. If the patient requires the drain to remain at time of discharge, the patient is fully instructed on drain care, emptying, and recording. The patient is then seen in the outpatient clinic, typically at approximately 7 after the surgery, the drain is removed regardless of output.

A standardized physical exam will be performed on all patients every day of inpatient stay by the chief resident and on postoperative appointment (5-8 days post-operatively) by the attending surgeon to evaluate for clinical evidence of seroma and hematomas.

Physical exam will specifically include:

1. Inspect and palpate for presence fluctuance.
2. Inspect for color change, erythema or ecchymosis
3. Palpate for tenderness

All patients will be given a patient satisfaction questionnaire at their first postoperative visit to evaluate their overall satisfaction with their hospital stay, their recovery and healing of their wound, their comfort with home care, and level of pain. The validated questionnaire, the measurement of quality of recovery (QoR-40), will be used.

Primary Endpoints and Outcomes

The primary outcome analyzed in this study will be total drain output (mL) in an effort to determine if the addition of Arista to the wound bed decreases overall wound drainage and drain output. Given that drain output influences time of drain removal, assessment will be made to determine if timing of drain removal differs between groups.

Secondary Endpoints

Secondary outcomes will allow for a robust analysis and will include:

1. Development of hematoma.
2. Development of seroma.
3. Requirement of patient to be discharged with drain.
4. Hospital length of stay.
5. Need for any additional procedures secondary wound complications.
6. The quantitative outcome from the patient satisfaction questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Total Thyroidectomy with or without lateral neck dissection
* Patient must be 18 years of age or older.
* The patient must have capacity to be able to sign a study-specific informed consent prior to study

Exclusion Criteria:

* Pregnancy (for female patients).
* Patients who will require anticoagulant medications other than routine DVT prophylaxis within 8 days postoperatively.
* Presence of clotting or bleeding disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Drain output | 1-14 days after Surgery
  Measured output from closed suction drain in ml. This will be recorded every 12 hrs until drain is removed.

SECONDARY OUTCOMES:
Seroma (Rate of clinically relevant seroma complications) | 1-14 days after surgery
  The rate of clinically relevant seroma complications will be evaluated for each group. Relevant seromas are those requiring intervention

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Mission Bay, San Francisco, California, United States